CLINICAL TRIAL: NCT05591118
Title: Pulmonary Embolism - Thrombus Removal With Catheter-Directed Therapy
Acronym: PE-TRACT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-01272
Record Dates: First submitted 2022-10-18; First posted 2022-10-24 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Embolism
Keywords: Catheter-Directed Therapy (CDT)
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Catheter-Directed Therapy (CDT) plus Anticoagulation (Experimental): Participants will receive CDT consisting of mechanical thrombectomy (MT) or intrathrombus catheter-directed thrombolysis (CDL) using FDA-cleared devices for pulmonary embolism (PE). The exact technique and devices used will be at the discretion of the endovascular physician, within parameters defined by the PE-TRACT Manual of Operations (MOP) and accepted standard care. Before and after CDT, patients will receive standard PE therapy as in the no-CDT Arm.
  Interventions: Drug: Anticoagulant Therapy; Device: Catheter-Directed Therapy
- No Catheter-Directed Therapy (No-CDT) (Active Comparator): Standard anticoagulant therapy (FDA-approved regimen) for the treatment of PE.
  Interventions: Drug: Anticoagulant Therapy

INTERVENTIONS:
Drug: Anticoagulant Therapy — All subjects will receive anticoagulation for a minimum of 3 months.
Device: Catheter-Directed Therapy — The endovascular physician can choose to use either mechanical thrombectomy (MT) using a device cleared by the FDA to treat PE or catheter-directed thrombolysis (CDL) using an infusion catheter cleared by the FDA to administer thrombolytic drugs for the treatment of PE
  Arms: Catheter-Directed Therapy (CDT) plus Anticoagulation

SUMMARY:
PE-TRACT is an open-label, assessor-blinded, randomized trial, aiming to compare catheter-directed therapy (CDT) and anticoagulation (CDT group) with anticoagulation alone (No-CDT) in 500 patients with submassive PE, proximal pulmonary artery thrombus and right ventricular dilation.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic PE diagnosed by contrast-enhanced CT angiography with involvement of a main or lobar pulmonary artery branch; and
2. Right ventricular (RV) dilation as defined by the presence of an RV/Left ventricular ratio > 1 on CT angiography

Exclusion Criteria:

1. Age < 18 years
2. Systolic blood pressure < 90 mmHg for >15 consecutive minutes or > 40 mmHg drop from baseline, or vasopressor requirement for blood pressure support (i.e., massive PE), occurring within 1 hour prior to eligibility assessment.
3. Symptom duration > 14 days for the current PE episode
4. Irreversible INR > 3
5. Irreversible Thrombocytopenia (Platelets < 50,000/microliter)
6. Creatinine > 2.0 mg/dl
7. Hemoglobin < 7.0 g/dl
8. Pregnancy (positive urine or blood pregnancy test (a pregnancy test must be obtained within 7 days prior to randomization in people of childbearing potential))
9. Allergy or hypersensitivity to Recombinant Tissue Plasminogen Activator (rt-PA), or iodinated contrast, except for mild-moderate contrast allergies for which steroid pre-medication can be used
10. Life expectancy < 1 year
11. Chronic inability to independently walk prior to the current PE episode (e.g. wheelchair dependent, walker or cane dependent, paraplegic, and/or bed-bound)
12. Allergy to heparin or history of Heparin-Induced Thrombocytopenia (HIT)
13. Unable or unwilling to provide informed consent
14. Major contraindication or unsuitability for all CDT methods available at the Clinical Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2027-03-29 (Estimated); Study Completion 2027-06-26 (Estimated)

PRIMARY OUTCOMES:
Peak Oxygen Consumption (PVO2) | Month 3
  PVO2 measured during cardiopulmonary exercise test (CPET).
New York Heart Association (NYHA) Functional Classification | Month 12
  The NYHA classifies the extent of heart failure. It classifies patients in one of four categories based on their limitations during physical activity; the limitations/symptoms are in regards to normal breathing and varying degrees in shortness of breath and or angina pain:
  * Class I - No symptoms and no limitation with ordinary physical activity.
  * Class II - Mild symptoms and slight limitation during ordinary activity.
  * Class III - Moderate limitation in activity (even less than ordinary) due to symptoms.
  * Class IV - Symptoms occur at rest and severe limitation with any physical activity.
  * Class V - Dead.
Incidence of Major Bleeding at Day 7 | Up to Day 7
  International Society on Thrombosis and Haemostasis (ISTH) definition of "Major Bleeding" to be used. Per ISTH, Major Bleeding defined as:
  1. Fatal bleeding, AND/OR;
  2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome, AND/OR;
  3. Bleeding causing a fall in hemoglobin level of 2 g/dL (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells.

SECONDARY OUTCOMES:
Six-Minute Walk Distance (6MWD) | Month 12
Short-Form Health Survey-36 (SF-36) Score | Month 12
  36-item questionnaire assessing general health. It measures 8 dimensions of health status: social function, physical function, emotional role, physical role, mental health, vitality, physical pain, and general health. Scores range from 0 (worst health status) to 100 (best health status).
Incidence of Clinical Deterioration (Fatal and Non-Fatal) at Day 7 | Up to Day 7
  Clinical deterioration defined as hemodynamic decompensation or respiratory decompensation requiring endotracheal intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Rao, MD, Principal Investigator — NYU Langone Health
Locations (40):
- United States (40):
  - The University of Alabama At Birmingham, Birmingham, Alabama
  - Stanford Medicine, Palo Alto, California
  - UC Davis Health, Sacramento, California
  - Scripps Memorial Hospital, La Jolla, San Diego, California
  - The Lundquist Institute, Torrance, California
  - Christiana Care, Newark, Delaware
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - Baptist Health Miami Cardiac & Vascular Institute, Miami, Florida
  - University of South Florida/ Tampa General Hospital, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Loyola University Chicago, Maywood, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - University of Iowa, Iowa City, Iowa
  - MaineHealth, Portland, Maine
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Trinity Health - Ann Arbor Hospital, Ypsilanti, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - NYU Langone Health - Tisch Hospital, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Promedica, Toledo, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Main Line Healh, Wynnewood, Pennsylvania
  - Lifespan, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Intermountain Health, Murray, Utah
  - University of Utah Health, Salt Lake City, Utah
  - Sentara Health Research Center, Norfolk, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: aks9010@med.cornell.edu.The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to aks9010@med.cornell.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Sista AK, Troxel AB, Tarpey T, Parpia S, Goldhaber SZ, Stringer WW, Magnuson EA, Cohen DJ, Kahn SR, Rao SV, Morris TA, Goldfeld KS, Vedantham S. Rationale and design of the PE-TRACT trial: A multicenter randomized trial to evaluate catheter-directed therapy for the treatment of intermediate-risk pulmonary embolism. Am Heart J. 2025 Mar;281:112-122. doi: 10.1016/j.ahj.2024.11.016. Epub 2024 Dec 3. PMID 39638275